CLINICAL TRIAL: NCT01693562
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI4736 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1/2 Study to Evaluate MEDI4736
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI4736-1108
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (23):
- Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) (Experimental): Participants will receive intravenous (IV) infusion of MEDI4736 (durvalumab) 0.1 mg/kg every 2 weeks (Q2W) in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) (Experimental): Participants will receive IV infusion of MEDI4736 0.3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Escalation Cohort (MEDI4736 1 mg/kg Q2W) (Experimental): Participants will receive IV infusion of MEDI4736 1 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Escalation Cohort (MEDI4736 3 mg/kg Q2W) (Experimental): Participants will receive IV infusion of MEDI4736 3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Escalation Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Escalation Cohort (MEDI4736 15 mg/kg Q3W) (Experimental): Participants will receive IV infusion of MEDI4736 15 mg/kg every 3 weeks (Q3W) in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Exploration Durvalumab 20 mg/kg (Q4W) (Experimental): Participants will receive IV infusion of MEDI4736 20 mg/kg every 4 weeks (Q4W) in the dose-exploration phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion Non-SCCHN Cohort HPV positive (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with non-SCCHN human papilloma virus positive (Non-SCCHN HPV+) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with non-small-cell lung cancer (NSCLC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with hepatocellular carcinoma (HCC Total) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with advance cutaneous melanoma (ACM) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with uveal melanoma (UM) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with gastroesophageal cancer (GEC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with triple-negative breast cancer (TNBC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with pancreatic adenocarcinoma (PAC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with urothelial carcinoma (UC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with glioblastoma multiforme (GBM) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose- expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with ovarian cancer (OC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with soft- tissue sarcoma (STS) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with small-cell lung cancer (SCLC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with microsatellite instability (MSI)-high cancer will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736
- Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W) (Experimental): Participants with nasopharyngeal carcinoma (NPC) will receive IV infusion of MEDI4736 10 mg/kg Q2W in the dose- expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736 — Participants will receive IV infusion of MEDI4736 for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Other Names: Durvalumab

SUMMARY:
This is a multicenter, open-label, first-time-in-human study with a standard 3+3 dose-escalation phase in participants with advanced solid tumors followed by an expansion phase in participants with advanced solid tumors. An exploration cohort has been added to determine the safety using every 4 weeks (Q4W) dosing.

DETAILED DESCRIPTION:
A dose-escalation and dose-expansion study of MEDI4736 (a monoclonal antibody that targets programmed cell death ligand-1 (PD-L1)) will evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity (IM), and antitumor activity of MEDI4736 in adult participants with solid tumors. A dose exploration cohort will look at the safety profile of Q4W dosing of MEDI4736.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* In the dose-escalation phase: histologically- or cytologically- confirmed advanced solid tumor that is refractory to standard therapy and for which no standard therapy exists.
* In the dose-expansion phase: histologically- or cytologically- confirmed advanced solid tumor where if an approved first-line therapy is available, participants must have failed, be intolerant to, be ineligible for, or have refused
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
* Adequate organ and marrow function.
* Participants must have at least 1 measurable lesion.
* Available archived tumor tissue sample.
* Willingness to provide consent for biopsy sample (dose-expansion only)

Exclusion Criteria:

* Any prior Grade ≥ 3 immune-mediated adverse event (imAE) while receiving immunotherapy
* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
* Prior treatment with immunotherapy agents including, but not limited to, tumor necrosis factor receptor superfamily agonists or checkpoint inhibitors or natural killer (NK) cell inhibitors.
* Active or prior documented autoimmune disease within the past 2 years
* History of primary immunodeficiency
* History of organ transplant that requires use of immunosuppressives
* Symptomatic or untreated central nervous system (CNS) metastases requiring concurrent treatment
* Other invasive malignancy within 2 years
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness
* Known history of tuberculosis
* Known to be human immunodeficiency virus (HIV) positive
* Known to be Hepatitis B or C positive (except HCC participants)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2012-09-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC — MedImmune LLC
Locations (71):
- United States (44):
  - Research Site, Scottsdale, Arizona
  - Research Site, Burbank, California
  - Research Site, Gilroy, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Whittier, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Hackensack, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Blacksburg, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
- Belgium (4):
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
- Canada (3):
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (2):
  - Research Site, Paris
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Berlin
  - Research Site, Gauting
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Minden
- Italy (4):
  - Research Site, Lecce
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Siena
- South Korea (4):
  - Research Site, Gwangju
  - Research Site, Seogu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (3):
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Sutton

REFERENCES:
- [Derived] Li Q, Cristini V, Gupta A, Achour I, Barrett JC, Koay EJ. Clinical Validation of Mathematically Derived Early Tumor Dynamics for Solid Tumors in Response to Durvalumab. JCO Clin Cancer Inform. 2024 Jul;8:e2300254. doi: 10.1200/CCI.23.00254. PMID 38996196
- [Derived] Gavrilov S, Zhudenkov K, Helmlinger G, Dunyak J, Peskov K, Aksenov S. Longitudinal Tumor Size and Neutrophil-to-Lymphocyte Ratio Are Prognostic Biomarkers for Overall Survival in Patients With Advanced Non-Small Cell Lung Cancer Treated With Durvalumab. CPT Pharmacometrics Syst Pharmacol. 2021 Jan;10(1):67-74. doi: 10.1002/psp4.12578. Epub 2020 Dec 21. PMID 33319498
- [Derived] Sheth S, Gao C, Mueller N, Angra N, Gupta A, Germa C, Martinez P, Soria JC. Durvalumab activity in previously treated patients who stopped durvalumab without disease progression. J Immunother Cancer. 2020 Aug;8(2):e000650. doi: 10.1136/jitc-2020-000650. PMID 32847985
- [Derived] Zhang Q, Luo J, Wu S, Si H, Gao C, Xu W, Abdullah SE, Higgs BW, Dennis PA, van der Heijden MS, Segal NH, Chaft JE, Hembrough T, Barrett JC, Hellmann MD. Prognostic and Predictive Impact of Circulating Tumor DNA in Patients with Advanced Cancers Treated with Immune Checkpoint Blockade. Cancer Discov. 2020 Dec;10(12):1842-1853. doi: 10.1158/2159-8290.CD-20-0047. Epub 2020 Aug 14. PMID 32816849
- [Derived] Zajac M, Ye J, Mukhopadhyay P, Jin X, Ben Y, Antal J, Gupta AK, Rebelatto MC, Williams JA, Walker J. Optimal PD-L1-high cutoff for association with overall survival in patients with urothelial cancer treated with durvalumab monotherapy. PLoS One. 2020 Apr 27;15(4):e0231936. doi: 10.1371/journal.pone.0231936. eCollection 2020. PMID 32339189
- [Derived] Nordstrom BL, Oguz M, Chu BC, Ouwens M, Arkenau HT, Klein AB. Effectiveness of durvalumab versus chemotherapy in metastatic urothelial cancer: an observational, indirect comparison. J Comp Eff Res. 2020 Feb;9(3):191-199. doi: 10.2217/cer-2019-0163. Epub 2020 Jan 9. PMID 31916448
- [Derived] Antonia SJ, Balmanoukian A, Brahmer J, Ou SI, Hellmann MD, Kim SW, Ahn MJ, Kim DW, Gutierrez M, Liu SV, Schoffski P, Jager D, Jamal R, Jerusalem G, Lutzky J, Nemunaitis J, Calabro L, Weiss J, Gadgeel S, Bhosle J, Ascierto PA, Rebelatto MC, Narwal R, Liang M, Xiao F, Antal J, Abdullah S, Angra N, Gupta AK, Khleif SN, Segal NH. Clinical Activity, Tolerability, and Long-Term Follow-Up of Durvalumab in Patients With Advanced NSCLC. J Thorac Oncol. 2019 Oct;14(10):1794-1806. doi: 10.1016/j.jtho.2019.06.010. Epub 2019 Jun 20. PMID 31228626
- [Derived] Althammer S, Tan TH, Spitzmuller A, Rognoni L, Wiestler T, Herz T, Widmaier M, Rebelatto MC, Kaplon H, Damotte D, Alifano M, Hammond SA, Dieu-Nosjean MC, Ranade K, Schmidt G, Higgs BW, Steele KE. Automated image analysis of NSCLC biopsies to predict response to anti-PD-L1 therapy. J Immunother Cancer. 2019 May 6;7(1):121. doi: 10.1186/s40425-019-0589-x. PMID 31060602
- [Derived] Segal NH, Ou SI, Balmanoukian A, Fury MG, Massarelli E, Brahmer JR, Weiss J, Schoffski P, Antonia SJ, Massard C, Zandberg DP, Khleif SN, Xiao F, Rebelatto MC, Steele KE, Robbins PB, Angra N, Song X, Abdullah S, Butler M. Safety and efficacy of durvalumab in patients with head and neck squamous cell carcinoma: results from a phase I/II expansion cohort. Eur J Cancer. 2019 Mar;109:154-161. doi: 10.1016/j.ejca.2018.12.029. Epub 2019 Feb 4. PMID 30731276
- [Derived] Zajac M, Boothman AM, Ben Y, Gupta A, Jin X, Mistry A, Sabalos C, Nielsen A, Manriquez G, Barker C, Antal J, Wang P, Patil P, Schechter N, Rebelatto MC, Walker J. Analytical Validation and Clinical Utility of an Immunohistochemical Programmed Death Ligand-1 Diagnostic Assay and Combined Tumor and Immune Cell Scoring Algorithm for Durvalumab in Urothelial Carcinoma. Arch Pathol Lab Med. 2019 Jun;143(6):722-731. doi: 10.5858/arpa.2017-0555-OA. Epub 2018 Nov 20. PMID 30457897
- [Derived] Steele KE, Tan TH, Korn R, Dacosta K, Brown C, Kuziora M, Zimmermann J, Laffin B, Widmaier M, Rognoni L, Cardenes R, Schneider K, Boutrin A, Martin P, Zha J, Wiestler T. Measuring multiple parameters of CD8+ tumor-infiltrating lymphocytes in human cancers by image analysis. J Immunother Cancer. 2018 Mar 6;6(1):20. doi: 10.1186/s40425-018-0326-x. PMID 29510739
- [Derived] Powles T, O'Donnell PH, Massard C, Arkenau HT, Friedlander TW, Hoimes CJ, Lee JL, Ong M, Sridhar SS, Vogelzang NJ, Fishman MN, Zhang J, Srinivas S, Parikh J, Antal J, Jin X, Gupta AK, Ben Y, Hahn NM. Efficacy and Safety of Durvalumab in Locally Advanced or Metastatic Urothelial Carcinoma: Updated Results From a Phase 1/2 Open-label Study. JAMA Oncol. 2017 Sep 14;3(9):e172411. doi: 10.1001/jamaoncol.2017.2411. Epub 2017 Sep 14. PMID 28817753
- [Derived] Levy A, Massard C, Soria JC, Deutsch E. Concurrent irradiation with the anti-programmed cell death ligand-1 immune checkpoint blocker durvalumab: Single centre subset analysis from a phase 1/2 trial. Eur J Cancer. 2016 Nov;68:156-162. doi: 10.1016/j.ejca.2016.09.013. Epub 2016 Oct 17. PMID 27764686
- See also: CSP amendment — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CD-ON-MEDI4736-1108&attachmentIdentifier=4cfe3393-2ef4-499b-af69-233e9ad1c75e&fileName=cd-on-medi4736-1108-csp-amendment-9-redacted_20201207.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CD-ON-MEDI4736-1108&attachmentIdentifier=b10f44de-43f5-4ffd-b0aa-5f4544600b45&fileName=cd-on-medi4736-1108-sap-ed-6-redacted_Redacted_20201207.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Belgium, Canada, France, Germany, Italy, South Korea, Taiwan, United Kingdom, and the United States of America.
Groups:
- Escalation Cohort (MEDI4736 0.1 mg/kg Q2W): Participants received intravenous (IV) infusion of MEDI4736 (durvalumab) 0.1 mg/kg every 2 weeks (Q2W) in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation Cohort (MEDI4736 0.3 mg/kg Q2W): Participants received IV infusion of MEDI4736 0.3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation Cohort (MEDI4736 1 mg/kg Q2W): Participants received IV infusion of MEDI4736 1 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation Cohort (MEDI4736 3 mg/kg Q2W): Participants received IV infusion of MEDI4736 3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation Cohort (MEDI4736 10 mg/kg Q2W): Participants received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation Cohort (MEDI4736 15 mg/kg Q3W): Participants received IV infusion of MEDI4736 15 mg/kg every 3 weeks (Q3W) in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Exploration Durvalumab 20 mg/kg (Q4W): Participants received IV infusion of MEDI4736 20 mg/kg every 4 weeks (Q4W) in the dose-exploration phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W): Participants with squamous cell carcinoma of the head and neck (SCCHN) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W): Participants with non-SCCHN human papilloma virus positive (Non-SCCHN HPV+) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W): Participants with non-small-cell lung cancer (NSCLC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W): Participants with hepatocellular carcinoma (HCC Total) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W): Participants with advance cutaneous melanoma (ACM) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion UM Cohort (MEDI4736 10 mg/kg Q2W): Participants with uveal melanoma (UM) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W): Participants with gastroesophageal cancer (GEC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W): Participants with triple-negative breast cancer (TNBC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W): Participants with pancreatic adenocarcinoma (PAC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion UC Cohort (MEDI4736 10 mg/kg Q2W): Participants with urothelial carcinoma (UC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W): Participants with glioblastoma multiforme (GBM) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose- expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion OC Cohort (MEDI4736 10 mg/kg Q2W): Participants with ovarian cancer (OC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion STS Cohort (MEDI4736 10 mg/kg Q2W): Participants with soft- tissue sarcoma (STS) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W): Participants with small-cell lung cancer (SCLC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W): Participants with microsatellite instability (MSI)-high cancer received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W): Participants with nasopharyngeal carcinoma (NPC) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose- expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Period: Escalation Phase
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Durvalumab 20 mg/kg (Q4W) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Started | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 2 | 0 | 3 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Exploration Phase
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Durvalumab 20 mg/kg (Q4W) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Durvalumab 20 mg/kg (Q4W) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 304 (2 eligible NSCLC participants from dose-escalation were added to the dose expansion summaries.) | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 300 | 40 | 21 | 23 | 51 | 40 | 31 | 197 | 20 | 47 | 20 | 21 | 62 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 2 | 54 | 2 | 2 | 3 | 5 | 16 | 7 | 40 | 4 | 8 | 3 | 1 | 8 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 42 | 17 | 208 | 30 | 8 | 19 | 42 | 23 | 23 | 128 | 16 | 36 | 16 | 17 | 35 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 10 | 4 | 4 | 1 | 3 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 28 | 4 | 7 | 0 | 1 | 1 | 0 | 28 | 0 | 1 | 0 | 1 | 17 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Durvalumab 20 mg/kg (Q4W) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W) | Total
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7 | 21 | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10 | 1024
Age, Customized [Count of Participants; unit: Participants] — Population: The data for this baseline measure is reported separately for each phase of the study.
  Participants
    Escalation Phase: number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27
    Escalation Phase: 18-64 years | 2 | 0 | 1 | 2 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Escalation Phase: 65-84 years | 2 | 4 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
    Escalation Phase: 85 years and above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Exploration Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Exploration Phase: 18-64 years | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
    Exploration Phase: 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Exploration Phase: 85 years and above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Expansion Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10 | 976
    Expansion Phase: 18-64 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 19 | 146 | 26 | 12 | 14 | 33 | 35 | 16 | 77 | 16 | 30 | 15 | 9 | 47 | 7 | 543
    Expansion Phase: 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 3 | 156 | 14 | 9 | 10 | 18 | 5 | 15 | 122 | 4 | 16 | 5 | 12 | 15 | 3 | 427
    Expansion Phase: 85 years and above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The data for this baseline measure is reported separately for each phase of the study.
  Participants
    Escalation Phase: number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27
    Escalation Phase: Female | 2 | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
    Escalation Phase: Male | 2 | 3 | 1 | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
    Exploration Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Exploration Phase: Female | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
    Exploration Phase: Male | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
    Expansion Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10 | 976
    Expansion Phase: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 15 | 133 | 8 | 9 | 10 | 13 | 40 | 9 | 58 | 7 | 47 | 15 | 8 | 34 | 3 | 418
    Expansion Phase: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 7 | 171 | 32 | 12 | 14 | 38 | 0 | 22 | 143 | 13 | 0 | 5 | 13 | 28 | 7 | 558
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The data for this baseline measure is reported separately for each phase of the study.
  Participants
    Escalation Phase: number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27
    Escalation Phase: Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Escalation Phase: Not Hispanic or Latino | 3 | 4 | 2 | 3 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23
    Escalation Phase: Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Exploration Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Exploration Phase: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Exploration Phase: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19
    Exploration Phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Expansion Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10 | 976
    Expansion Phase: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 12 | 2 | 2 | 1 | 4 | 0 | 1 | 5 | 2 | 2 | 5 | 1 | 4 | 0 | 47
    Expansion Phase: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 54 | 21 | 287 | 32 | 19 | 18 | 43 | 33 | 30 | 177 | 18 | 39 | 15 | 20 | 42 | 10 | 858
    Expansion Phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 6 | 0 | 5 | 4 | 7 | 0 | 19 | 0 | 6 | 0 | 0 | 16 | 0 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The data for this baseline measure is reported separately for each phase of the study.
  Participants
    Escalation Phase: number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27
    Escalation Phase: American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Escalation Phase: Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Escalation Phase: Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Escalation Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Escalation Phase: White | 4 | 3 | 2 | 2 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
    Escalation Phase: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Escalation Phase: Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Escalation Phase: Missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Exploration Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
    Exploration Phase: American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Exploration Phase: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Exploration Phase: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Exploration Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Exploration Phase: White | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19
    Exploration Phase: Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Exploration Phase: Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Exploration Phase: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Expansion Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10 | 976
    Expansion Phase: American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Expansion Phase: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 58 | 9 | 0 | 0 | 1 | 2 | 0 | 40 | 0 | 4 | 1 | 2 | 6 | 5 | 134
    Expansion Phase: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 10 | 3 | 1 | 0 | 1 | 6 | 1 | 8 | 0 | 1 | 1 | 1 | 2 | 0 | 38
    Expansion Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
    Expansion Phase: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 19 | 227 | 19 | 19 | 19 | 45 | 25 | 29 | 128 | 19 | 36 | 18 | 17 | 34 | 3 | 706
    Expansion Phase: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 0 | 0 | 1 | 4 | 0 | 20
    Expansion Phase: Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Expansion Phase: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 5 | 6 | 1 | 5 | 3 | 6 | 0 | 19 | 0 | 6 | 0 | 0 | 16 | 0 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities in the Dose-escalation Phase
Description: A DLT was defined as any Grade 3 or higher treatment-related toxicity that occurred during the DLT-evaluation period including any >= Grade 3 colitis or >= Grade 3 immune-related adverse event (irAE; AEs of immune nature in the absence of a clear alternative etiology) including rash, pruritus, or diarrhea that did not downgrade to =< Grade 2 within 3 days after onset of the event despite maximal supportive care including systemic corticosteroids. The DLT-evaluation period for 0.1 to 10 mg/kg arms was from Day 1 to Day 28 of first dose and for 15 mg/kg arm was from Day 1 to Day 42 of first dose.
Time Frame: For MEDI4736 0.1 to MEDI4736 10 mg/kg arms: from Day 1 to Day 28 of first dose; for MEDI4736 15 mg/kg arm: from Day 1 to Day 42 of first dose
Population: DLT-evaluable population included all participants in the dose-escalation phase who received at least 2 doses of study drug and completed safety follow-up through DLT-evaluable period or experienced any DLT during the DLT-evaluation period.
Measure: Count of Participants; unit: Participants
Groups:
- Escalation Cohort (MEDI4736 0.3 mg/kg Q2W): Participants received IV infusion of MEDI4736 0.3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation , whichever occurred first
- Escalation Cohort (MEDI4736 3 mg/kg Q2W): Participants received IV infusion of MEDI4736 3 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation , whichever occurred first.
- Escalation Cohort (MEDI4736 10 mg/kg Q2W): Participants received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-escalation phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation , whichever occurred first.
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) in the Dose-escalation, Dose-exploration, and Dose-expansion Phase
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From Day 1 through 90 days after the last dose of study drug (approximately 5.25 years)
Population: As-treated population included all participants who received any dose of study drug. Participants enrolled in the 10 mg/kg Q2W Expansion and Escalation Cohort have been summarized as a total only. This is because the safety profile of durvalumab monotherapy 10 mg/kg Q2W was manageable and generally consistent with the known safety profile of the anti-programmed cell death ligand (PD-L1/PD-1) drug class.
Measure: Count of Participants; unit: Participants
Groups:
- Exploration Cohort (MEDI4736 20 mg/kg Q4W): Participants received IV infusion of MEDI4736 20 mg/kg every 4 weeks (Q4W) in the dose-exploration phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Escalation/Expansion Cohort (Total MEDI4736 10 mg/kg Q2W): Participants received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-escalation or dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation , whichever occurred first.
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W) | Escalation/Expansion Cohort (Total MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 21 | 980
Participants
  Any TEAEs | 3 | 4 | 3 | 3 | 7 | 21 | 963
  Any TESAEs | 1 | 2 | 1 | 1 | 3 | 13 | 536

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in the Dose-escalation, Dose-exploration, and Dose-expansion Phase
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of coagulation, urine, hematology, and serum chemistry.
Time Frame: From Day 1 through 90 days after the last dose of study drug (approximately 5.25 years)
Population: As-treated population included all participants who received any dose of study drug. Participants enrolled in the 10 mg/kg Q2W Expansion and Escalation Cohort have been summarized as a total only. This is because the safety profile of durvalumab monotherapy 10 mg/kg Q2W was manageable and generally consistent with the known safety profile of the anti-PD-L1/PD-1 drug class.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W) | Escalation/Expansion Cohort (Total MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 21 | 980
Participants
  Anaemia | 1 | 0 | 0 | 0 | 0 | 0 | 166
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 1 | 24
  White blood cell count increased | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 20
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 12
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Thrombocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Iron deficiency anaemia | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Haemoglobin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Neutrophil count increased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Red blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Anaemia of chronic disease | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Eosinophilia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Haemolysis | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leukostasis syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Immune thrombocytopenic purpura | 0 | 0 | 0 | 0 | 0 | 0 | 1
  International normalised ratio increased | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 15
  Blood fibrinogen increased | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Disseminated intravascular coagulation | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Prothrombin time prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Activated partial thromboplastin time shortened | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Coagulation factor increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Coagulopathy | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 1 | 0 | 1 | 2 | 77
  Aspartate aminotransferase increased | 0 | 0 | 1 | 0 | 1 | 2 | 99
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 | 1 | 70
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 1 | 42
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 0 | 2 | 71
  Hyperbilirubinaemia | 0 | 0 | 0 | 0 | 0 | 0 | 14
  Transaminases increased | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Hepatic function abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Alanine aminotransferase decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood albumin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hepatic enzyme increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Liver function test increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Blood creatinine increased | 0 | 1 | 1 | 0 | 0 | 0 | 46
  Hyperuricaemia | 0 | 0 | 0 | 0 | 0 | 0 | 22
  Blood urea increased | 0 | 0 | 0 | 0 | 0 | 0 | 10
  Glomerular filtration rate decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hypothyroidism | 0 | 1 | 1 | 0 | 1 | 3 | 89
  Hyperthyroidism | 0 | 0 | 0 | 0 | 0 | 1 | 30
  Blood thyroid stimulating hormone increased | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Blood thyroid stimulating hormone decreased | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Thyroxine decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Thyroxine free decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Thyroxine free increased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Tri-iodothyronine free decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Thyroxine increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Tri-iodothyronine decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Tri-iodothyronine increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyponatraemia | 0 | 0 | 1 | 0 | 1 | 1 | 91
  Hypomagnesaemia | 0 | 0 | 0 | 0 | 0 | 1 | 55
  Hypercalcaemia | 0 | 0 | 0 | 0 | 0 | 0 | 47
  Hyperglycaemia | 0 | 0 | 1 | 0 | 0 | 0 | 32
  Hypokalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 60
  Hypocalcaemia | 0 | 0 | 0 | 0 | 0 | 0 | 17
  Hypophosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Hypertriglyceridaemia | 0 | 0 | 0 | 0 | 0 | 0 | 13
  Hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 0 | 10
  Blood cholesterol increased | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Blood magnesium decreased | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Blood triglycerides increased | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Blood glucose increased | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Hypercholesterolaemia | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Blood potassium increased | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Blood chloride increased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood electrolytes decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood potassium decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Protein total decreased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Protein urine present | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood bicarbonate decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood chloride decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood sodium decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypermagnesaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypernatraemia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypochloraemia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoproteinaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyperkalaemia | 0 | 0 | 0 | 0 | 0 | 0 | 30

4. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs in the Dose-escalation, Dose-exploration, and Dose-expansion Phase
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (body weight, body temperature, blood pressure, pulse rate, and respiratory rate).
Time Frame: From Day 1 through 90 days after the last dose of study drug (approximately 5.25 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W) | Escalation/Expansion Cohort (Total MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 21 | 980
Participants
  Pyrexia | 0 | 3 | 0 | 1 | 3 | 2 | 145
  Weight decreased | 0 | 0 | 0 | 0 | 0 | 2 | 79
  Hypertension | 0 | 1 | 0 | 1 | 0 | 0 | 31
  Hypotension | 0 | 0 | 0 | 0 | 0 | 1 | 36
  Weight increased | 0 | 0 | 0 | 0 | 0 | 0 | 22
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 19
  Sinus tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 14
  Arrhythmia | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Sinus bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Heart rate increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Heart rate irregular | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Peak expiratory flow rate decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Change From Baseline in QT/QTc Interval in Local Electrocardiogram in the Dose-escalation, Dose-exploration, and Dose-expansion Phase
Description: Number of participants with change from baseline in notable QT/QTc interval in local electrocardiogram (ECG) are reported. The data for >0 participants with notable QT/QTc interval in local ECG from baseline are reported.
Time Frame: From Baseline (Day 1) through 90 days after the last dose of study drug (approximately 5.25 years)
Population: As-treated population included all participants who received any dose of study drug were analyzed. Participants with ECG readings available were evaluable for this analysis. Participants enrolled in the 10 mg/kg Q2W Expansion and Escalation Cohort have been summarized as a total only. This is because the safety profile of durvalumab monotherapy 10 mg/kg Q2W was manageable and generally consistent with the known safety profile of the anti-PD-L1/PD-1 drug class.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W) | Escalation/Expansion Cohort (Total MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 21 | 980
Participants
  QTcF: > 30 (msec): number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 63
  QTcF: > 30 (msec) |  | 1 | 0 | 0 |  |  | 4
  QTcF: > 60 (msec): number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 63
  QTcF: > 60 (msec) |  | 1 | 0 | 0 |  |  | 0
  QTcB: > 30 (msec): number analyzed (Participants) | 2 | 2 | 2 | 1 | 2 | 9 | 288
  QTcB: > 30 (msec) | 0 | 0 | 0 | 0 | 0 | 4 | 17
  QTcB: > 60 (msec): number analyzed (Participants) | 2 | 2 | 2 | 1 | 2 | 9 | 288
  QTcB: > 60 (msec) | 0 | 0 | 0 | 0 | 0 | 0 | 4
  QTcB: > 90 (msec): number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 21 | 288
  QTcB: > 90 (msec) | 0 | 0 | 0 | 0 | 0 | 0 | 3

6. Primary Outcome: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) in Participants With Non-squamous NSCLC Who Had Received 2 or More Prior Lines of Therapy in the Dose-expansion Phase
Description: The ORR assessed by BICR in participants with non-squamous NSCLC who had received 2 or more prior lines of therapy is reported. The ORR is defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1). The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as two CRs that were separated by at least 28 days with no evidence of progression in-between. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: From Day 1 through disease progression, study withdrawal, or initiation of another anticancer therapy, whichever occurred first (approximately 5.25 years)
Population: Participants with non-squamous NSCLC in Full analysis set (FAS) population who had received 2 or more prior line of therapy were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expansion Non-squamous NSCLC 3L+ Cohort: Participants with non-squamous NSCLC who had received 2 or more lines of prior therapy (3L+) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion Non-squamous NSCLC 3L+ Cohort
Number analyzed (Participants) | 68
Percentage of participants | 10.3 [4.2 to 20.1]

7. Primary Outcome: ORR Assessed by BICR in Participants With Squamous NSCLC Who Had Received 1 and 2 or More Prior Lines of Therapy in the Dose-expansion Phase
Description: The ORR assessed by BICR in participants with squamous NSCLC who had received 1 and 2 or more prior lines of therapy is reported. The ORR is defined as BOR of confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as two CRs that were separated by at least 28 days with no evidence of progression in-between. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 6
Population: Participants with squamous NSCLC in FAS population who had received 1 and 2 or more prior lines of therapy were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expansion Squamous NSCLC 2L+ Cohort: Participants with squamous NSCLC who had received at least 1 line of prior therapy (2L+) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion Squamous NSCLC 3L+ Cohort: Participants with squamous NSCLC who had received 2 or more lines of prior therapy (3L+) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion Squamous NSCLC 2L+ Cohort | Expansion Squamous NSCLC 3L+ Cohort
Number analyzed (Participants) | 117 | 62
Percentage of participants | 12.8 [7.4 to 20.3] | 12.9 [5.7 to 23.9]

8. Primary Outcome: ORR Assessed by BICR in Participants With UC Post-platinum (Programmed Cell Death Ligand [PD-L1] Status High) Who Had Received at Least 1 Line of Prior Therapy (2L+) in the Dose-expansion Phase
Description: The ORR assessed by BICR in participants with UC post-platinum PD-L1 status high 2L+ is reported. The ORR is defined as BOR of confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as two CRs that were separated by at least 28 days with no evidence of progression in-between. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 6
Population: Participants with UC in FAS population with 2L+ post-platinum PD-L1 status high (>= 25% tumor cell membrane or >= 25% immune cell staining) were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expansion UC PD-L1 High 2L+ Cohort: Participants with UC (post-platinum PD-L1 status high) who had received at least 1 line of prior therapy (2L+) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion UC PD-L1 High 2L+ Cohort
Number analyzed (Participants) | 98
Percentage of participants | 27.6 [19.0 to 37.5]

9. Secondary Outcome: Area Under the Serum Concentration-time Curve up to the Last Measurable Concentration (AUClast) of MEDI4736 After the First Dose in the Dose-escalation and Dose-exploration Phase
Description: Area under the concentration-time curve from time zero to the last measurable concentration (AUClast) of MEDI4736 is reported.
Time Frame: After the first dose between Day 0 and Day 15 (Day 1 [pre and post dose] and predose of Dose 2 for all cohorts; Days 3, 5, 10 for Cohorts 0.1mg/kg to 10 mg/kg; Days 3, 5, 10, 15 for Cohort 15 mg/kg; Day 15 for Cohort 20 mg/kg)
Population: Pharmacokinetics (PK) evaluable population included all participants who received any dose of study drug and had at least one postdose PK concentration. Non-compartmental PK analysis was conducted using the data from dose escalation and exploration phases only. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*µg/mL
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 5 | 7 | 18
Day*µg/mL | 5.144 (45.1) | 25.063 (65.5) | 130.546 (20.1) | 399.863 (21.7) | 1780.152 (39.1) | 2943.770 (36.3) | 4501.888 (23.1)

10. Secondary Outcome: Maximum Serum Concentration (Cmax) of MEDI4736 After the First Dose in the Dose-escalation and Dose-exploration Phase
Description: The Cmax of MEDI4736 is reported.
Time Frame: as for outcome 9
Population: The PK evaluable population included all participants who received any dose of study drug and had at least one postdose PK concentration. Non-compartmental PK analysis was conducted using the data from dose escalation and exploration phases only. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Cohort (MEDI4736 20 mg/kg Q4W)
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 5 | 7 | 18
µg/mL | 2.780 (22.1) | 7.969 (23.0) | 22.773 (11.3) | 70.807 (17.0) | 293.540 (23.4) | 427.085 (25.5) | 416.051 (23.9)

11. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI4736 in the Dose-escalation, Dose-exploration Phase, and Dose-expansion Phase.
Description: Number of participants with positive ADA titer to MEDI4736 are reported. Treatment-boosted ADA is defined as baseline positive ADA titer that was boosted to a 4-fold or higher level following drug administration; persistent positive is defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment; and transient positive is defined as having at least one post-baseline ADA-positive assessment and not fulfilling the condition of persistent positive.
Time Frame: Escalation: Day1 of Dose(D)1 & D3, even numbered doses after D4; Exploration: Day1 of D1 & D2, even numbered doses after D2; Expansion: Day1 of D1, every 12 weeks since D3; all phases: till EOT, 30 days and 3 and 6 months post last dose (~5.25 years)
Population: The ADA evaluable population included all participants who received any dose of study drug, had non-missing baseline (before Day 1) ADA, and at least one non-missing post-baseline ADA results. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Total Escalation/Exploration Cohort: Participants received IV infusion of MEDI4736 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg Q2W, and 15 mg/kg Q3W in the dose-escalation phase; and 20 mg/kg every 4 weeks (Q4W) in the dose-exploration phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Total Escalation/Exploration Cohort | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 45 | 56 | 17 | 257 | 37 | 17 | 21 | 38 | 33 | 26 | 148 | 17 | 41 | 19 | 15 | 58 | 6
Participants
  Positive post-baseline | 4 | 1 | 0 | 6 | 0 | 0 | 1 | 0 | 1 | 0 | 7 | 0 | 2 | 1 | 0 | 2 | 0
  Treatment-boosted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Persistent positive | 2 | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 0 | 0 | 1 | 0 | 1 | 0
  Transient positive | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0

12. Secondary Outcome: Number of Participants With Best Overall Response (BOR) Assessed by BICR in NSCLC and SCCHN Cohort in the Dose-expansion Phase
Description: The BOR assessed by BICR based on RECIST v1.1 in NSCLC and SCCHN cohorts is reported. The BOR includes CR, PR, stable disease (SD), progressive disease (PD), and non-evaluable (NE). The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. The PD is defined at least 20% increase in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The NE is defined as either when no or only a subset of lesion measurements are made at an assessment.
Time Frame: as for outcome 6
Population: Participants in FAS population with NSCLC and SCCHN were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Count of Participants; unit: Participants
Groups:
- Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W): Participants with SCCHN received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W): Participants with NSCLC received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 55 | 275
Participants
  CR | 0 | 3
  PR | 4 | 39
  SD | 10 | 80
  PD | 31 | 110
  NE | 10 | 43

13. Secondary Outcome: Number of Participants With BOR Assessed by Investigator in the Dose-escalation, Dose-exploration, and Dose-expansion Phase
Description: The BOR assessed by investigator based on RECIST v1.1 is reported. The BOR includes CR, PR, SD, PD, and NE. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. The PD is defined at least 20% increase in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The NE is defined as either when no or only a subset of lesion measurements are made at an assessment.
Time Frame: as for outcome 6
Population: As-treated population included all participants who received any dose of study drug. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure. One participant from non-SCCHN HPV positive cohort had non-evaluable disease at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Total Escalation/Exploration Cohort: Participants received IV infusion of MEDI4736 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg Q2W, and 15 mg/kg Q3W in the dose-escalation phase; and 20 mg/kg Q4W in the dose-exploration phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Total Escalation/Exploration Cohort | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 48 | 62 | 22 | 302 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10
Participants
  CR | 1 | 1 | 1 | 5 | 0 | 1 | 0 | 1 | 0 | 0 | 18 | 0 | 1 | 0 | 0 | 3 | 0
  PR | 4 | 6 | 2 | 49 | 4 | 2 | 1 | 1 | 1 | 1 | 24 | 0 | 2 | 2 | 2 | 12 | 3
  SD | 18 | 14 | 7 | 102 | 22 | 9 | 8 | 17 | 8 | 6 | 45 | 5 | 18 | 8 | 4 | 27 | 2
  PD | 18 | 33 | 9 | 103 | 12 | 5 | 12 | 21 | 25 | 17 | 81 | 14 | 22 | 8 | 9 | 15 | 3
  NE | 7 | 8 | 2 | 43 | 2 | 4 | 3 | 11 | 6 | 7 | 33 | 1 | 4 | 2 | 6 | 5 | 2
  Not applicable | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Duration of Response (DoR) Assessed by BICR in NSCLC and SCCHN Cohort in the Dose-expansion Phase
Description: The DoR assessed by BICR in NSCLC and SCCHN cohorts is reported. The DoR is defined as the duration from the first documentation of objective response (OR) (confirmed CR or confirmed PR) to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between. The DoR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: Participants in FAS population with NSCLC and SCCHN were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017. The DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W): Participants with squamous SCCHN received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 4 | 42
Months | 12.37 [3.5 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 17.74 [5.6 to 38.0]

15. Secondary Outcome: DoR Assessed by Investigator in the Dose-expansion Phase
Description: The DoR in participants assessed by the investigator is reported. The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between. The DoR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: As-treated population included all participants who received any dose of study drug. The DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 7 | 3 | 54 | 4 | 3 | 1 | 2 | 1 | 1 | 42 | 0 | 3 | 2 | 2 | 15 | 3
Months | 19.71 [1.9 to 44.0] | 14.75 [12.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 9.95 [8.3 to 16.4] | 16.20 [7.2 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [7.9 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 9.23 [NA to NA] — 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [NA to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [NA to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 5.36 [NA to NA] — 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [14.6 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. |  | 24.87 [4.8 to 24.9] | 7.92 [6.1 to 9.7] | 23.51 [14.6 to 32.4] | 26.91 [12.7 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 8.64 [4.4 to 16.3]

16. Secondary Outcome: Disease Control Rate (DCR) Assessed by BICR in NSCLC and SCCHN Cohort in the Dose-expansion Phase
Description: Percentage of participants with disease control assessed by BICR in NSCLC and SCCHN cohorts is reported. Disease control is defined as a BOR of confirmed CR, confirmed PR, or SD based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: as for outcome 6
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 55 | 275
Percentage of participants | 25.5 [14.7 to 39.0] | 44.4 [38.4 to 50.5]

17. Secondary Outcome: DCR Assessed by Investigator in the Dose-expansion Phase
Description: Percentage of participants with disease control assessed by the investigator is reported. Disease control is defined as a BOR of confirmed CR, confirmed PR, or SD based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: as for outcome 6
Population: As-treated population included all participants who received any dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 62 | 22 | 302 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10
Percentage of participants | 33.9 [22.3 to 47.0] | 45.5 [25.7 to 70.2] | 51.7 [45.9 to 57.4] | 65.0 [48.3 to 79.4] | 57.1 [34.0 to 78.2] | 37.5 [18.8 to 59.4] | 37.3 [24.1 to 51.9] | 22.5 [10.8 to 38.5] | 22.6 [9.6 to 41.1] | 43.3 [36.3 to 50.4] | 0 [NA to NA] — 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 44.7 [30.2 to 59.9] | 50.0 [27.2 to 72.8] | 28.6 [11.3 to 52.2] | 67.7 [54.7 to 79.1] | 50.0 [18.7 to 81.3]

18. Secondary Outcome: Progression-free Survival (PFS) Assessed by BICR in NSCLC Cohort in the Dose-expansion Phase
Description: The PFS assessed by BICR in NSCLC cohort is reported. The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: Participants in As-treated population with NSCLC were analyzed. As-treated population included all participants who received any dose of study drug.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 304
Percentage of participants | 2.1 [1.5 to 2.6]

19. Secondary Outcome: PFS Assessed by BICR in SCCHN Cohort in the Dose-expansion Phase
Description: The PFS assessed by BICR in SCCHN cohort is reported. The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: Participants in FAS population with SCCHN were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 62
Percentage of participants | 1.4 [1.3 to 1.5]

20. Secondary Outcome: PFS Assessed by Investigator in the Dose-expansion Phase
Description: The PFS assessed by the investigator is reported. The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: As-treated population included all participants who received any dose of study drug. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 62 | 22 | 302 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10
Months | 1.4 [1.4 to 1.6] | 1.5 [1.2 to 5.6] | 2.6 [1.9 to 3.2] | 2.7 [1.4 to 5.3] | 2.8 [1.2 to 9.1] | 1.4 [1.3 to 4.6] | 1.4 [1.2 to 2.4] | 1.3 [1.2 to 1.6] | 1.5 [1.3 to 1.7] | 1.8 [1.4 to 2.6] | 1.4 [1.2 to 2.3] | 1.8 [1.4 to 2.7] | 2.6 [1.4 to 3.0] | 1.5 [0.9 to 1.8] | 5.4 [2.9 to 11.1] | 2.2 [0.7 to 5.7]

21. Secondary Outcome: OS in the Dose-Expansion Phase
Description: OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
Number analyzed (Participants) | 62 | 22 | 304 | 40 | 21 | 24 | 51 | 40 | 31 | 201 | 20 | 47 | 20 | 21 | 62 | 10
Months | 8.4 [5.7 to 12.3] | 11.6 [3.0 to 22.8] | 12.4 [9.3 to 15.2] | 13.2 [6.3 to 23.0] | NA [15.1 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 8.4 [4.5 to 14.3] | 4.9 [2.6 to 9.1] | 5.5 [3.5 to 16.8] | 5.7 [4.8 to 8.0] | 10.5 [6.9 to 15.7] | 10.0 [6.2 to 13.0] | 11.1 [8.2 to 16.6] | 15.8 [8.1 to 23.3] | 4.8 [1.3 to 10.4] | 24.1 [12.4 to 37.1] | 16.1 [0.9 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

22. Secondary Outcome: ORR Assessed by BICR in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The ORR assessed by BICR in UC cohort is reported. The ORR is defined as confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as two CRs that were separated by at least 28 days with no evidence of progression in-between. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in the FAS population were analyzed. FAS population included all participnats who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expansion UC PD-L1 Low/Negative Cohort: Participants with UC (PD-L1 status low/Negative) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion UC Total Cohort: Participants with UC (Total PD-L1 status - high, low/Negative, and unknown) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
- Expansion UC PD-L1 High Cohort: Participants with UC (PD-L1 status high) received IV infusion of MEDI4736 10 mg/kg Q2W in the dose-expansion phase for maximum of 12 months or until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurred first.
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 85 | 199 | 101
Percentage of participants | 5.9 [1.9 to 13.2] | 17.6 [12.6 to 23.6] | 27.7 [19.3 to 37.5]

23. Secondary Outcome: ORR Assessed by Investigator in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The ORR assessed by the investigator in UC cohort is reported. The ORR is defined as confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. A confirmed CR is defined as two CRs that were separated by at least 28 days with no evidence of progression in-between. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in the As-treated population were analyzed. As-treated population included all participants who received any dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 86 | 201 | 102
Percentage of participants | 7.0 [2.6 to 14.6] | 20.9 [15.5 to 27.2] | 33.3 [24.3 to 43.4]

24. Secondary Outcome: DoR Assessed by BICR in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The DoR assessed by BICR in UC cohort is reported. The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between. The DoR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in FAS population (all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 wks by 16Oct2017) were analyzed. DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 5 | 35 | 28
Months | 12.25 [8.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [16.0 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [16.0 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

25. Secondary Outcome: DoR Assessed by Investigator in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The DoR assessed by investigator in UC cohort is reported. The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an un-confirmed CR that were separated by at least 4 weeks with no evidence of progression in-between. The DoR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in the As-treated population were analyzed. As-treated population included all participants who received any dose of study drug. The DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 6 | 42 | 34
Months | 14.82 [6.9 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 19.71 [14.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [12.3 to NA] — Median and Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

26. Secondary Outcome: DCR Assessed by BICR in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: Percentage of participants with disease control assessed by BICR in UC cohort is reported. The DCR is defined as a BOR of confirmed CR, confirmed PR, or SD based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in the FAS population were analyzed. FAS population included all participants who received any dose of study drug, had measurable disease at baseline (Day 1) per BICR and were followed for at least 24 weeks by 16Oct2017.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 85 | 199 | 101
Percentage of participants | 21.2 [13.1 to 31.4] | 35.2 [28.6 to 42.2] | 43.6 [33.7 to 53.8]

27. Secondary Outcome: DCR Assessed by Investigator in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: Percentage of participants with disease control assessed by investigator in UC cohort is reported. Disease control is defined as a best overall response of confirmed CR, confirmed PR, or SD based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 28 days with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR not sufficient increase to qualify for disease progression.
Time Frame: as for outcome 6
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 86 | 201 | 102
Percentage of participants | 30.2 [20.8 to 41.1] | 43.3 [36.3 to 50.4] | 53.9 [43.8 to 63.8]

28. Secondary Outcome: PFS Assessed by BICR in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The PFS assessed by BICR in UC cohort is reported. The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as low/negative (<25% tumor cell membrane and <25% immune cell staining), total (PD-L1 high, PD-L1 low/negative, and PD-L1 unknown), and high (>= 25% tumor cell membrane or >=25% immune cell staining) included in the As-treated population were analyzed. As-treated population included all participants who received any dose of study drug. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 86 | 201 | 102
Months | 1.4 [1.3 to 1.5] | 1.5 [1.4 to 1.8] | 1.9 [1.4 to 2.7]

29. Secondary Outcome: PFS Assessed by Investigator in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The PFS assessed by the investigator in UC cohort is reported. The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 86 | 201 | 102
Months | 1.4 [1.4 to 1.7] | 1.8 [1.4 to 2.6] | 2.8 [1.8 to 3.7]

30. Secondary Outcome: OS in UC Cohort (PD-L1 Low/Negative, Total, and PD-L1 High) in the Dose-expansion Phase
Description: The OS in UC cohort is reported. The OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 Low/Negative Cohort | Expansion UC Total Cohort | Expansion UC PD-L1 High Cohort
Number analyzed (Participants) | 86 | 201 | 102
Months | 4.8 [3.3 to 8.1] | 10.5 [6.9 to 15.7] | 19.8 [9.3 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

31. Secondary Outcome: Adjusted Comparison of PFS by PD-L1 Status in UC Cohort in the Dose-expansion Phase
Description: The PFS by PD-L1 status in UC cohort is reported. The PFS estimates are adjusted for baseline eastern cooperative oncology (ECOG), smoking status, race, gender, age, previous lines of therapy, and liver metastasis. 95% CIs based on log (-log(survival)). The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: The UC cohort participants with PD-L1 status as high (>= 25% tumor cell membrane or >=25% immune cell staining) and low/negative (<25% tumor cell membrane and <25% immune cell staining) included in the As-treated population were analyzed. As-treated population included all participants who received any dose of study drug. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 High Cohort | Expansion UC PD-L1 Low/Negative Cohort
Number analyzed (Participants) | 61 | 39
Months | 2.6 [1.4 to 3.9] | 1.5 [1.4 to 2.4]
Statistical Analysis 1: Comparison: Expansion UC PD-L1 High Cohort vs Expansion UC PD-L1 Low/Negative Cohort; Test type: Equivalence — Other; p = 0.016, Regression, Cox

32. Secondary Outcome: Adjusted Comparison of OS by PD-L1 Status in UC Cohort in the Dose-expansion Phase
Description: The OS by PD-L1 status in UC cohort is reported. The OS estimates are adjusted for baseline ECOG, smoking status, race, gender, age, previous lines of therapy, and liver metastasis. 95% CIs based on log (-log(survival)). The OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 6
Population: as for outcome 31
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion UC PD-L1 High Cohort | Expansion UC PD-L1 Low/Negative Cohort
Number analyzed (Participants) | 61 | 39
Months | 18.4 [7.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 3.4 [2.4 to 14.3]
Statistical Analysis 1: Comparison: Expansion UC PD-L1 High Cohort vs Expansion UC PD-L1 Low/Negative Cohort; Test type: Equivalence — Other; p = 0.0046, Regression, Cox

ADVERSE EVENTS:
Time Frame: From Day 1 through 90 days after the last dose of study drug (approximately 5.25 years)
Arm/Group | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) | Exploration Durvalumab 20 mg/kg (Q4W) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W)
All-Cause Mortality (participants affected / at risk) | 4/4 | 2/4 | 0/3 | 3/3 | 6/6 | 4/7 | 17/21 | 42/62 | 17/22 | 208/304 | 30/40 | 8/21 | 19/24 | 42/51 | 23/40 | 23/31 | 128/201 | 16/20 | 36/47 | 16/20 | 17/21 | 35/62 | 7/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 1/3 | 1/3 | 3/6 | 3/7 | 13/21 | 30/62 | 16/22 | 163/304 | 24/40 | 7/21 | 12/24 | 26/51 | 20/40 | 25/31 | 117/201 | 9/20 | 26/47 | 7/20 | 14/21 | 31/62 | 7/10
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 3/3 | 3/3 | 6/6 | 7/7 | 20/21 | 61/62 | 22/22 | 292/304 | 40/40 | 19/21 | 22/24 | 50/51 | 39/40 | 31/31 | 194/201 | 18/20 | 46/47 | 20/20 | 17/21 | 57/62 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) (N=4) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) (N=4) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) (N=3) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) (N=3) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) (N=6) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) (N=7) | Exploration Durvalumab 20 mg/kg (Q4W) (N=21) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) (N=62) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) (N=22) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) (N=304) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) (N=40) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) (N=21) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) (N=24) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) (N=51) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) (N=40) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) (N=31) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) (N=201) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) (N=20) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) (N=47) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) (N=20) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) (N=21) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) (N=62) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (5) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 7 (11) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 21 (29) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (10) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (13) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood electrolytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eastern cooperative oncology group performance status worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 45 (50) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 47 (55) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (13) | 0 (0) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 23 (24) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 3 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Cohort (MEDI4736 0.1 mg/kg Q2W) (N=4) | Escalation Cohort (MEDI4736 0.3 mg/kg Q2W) (N=4) | Escalation Cohort (MEDI4736 1 mg/kg Q2W) (N=3) | Escalation Cohort (MEDI4736 3 mg/kg Q2W) (N=3) | Escalation Cohort (MEDI4736 10 mg/kg Q2W) (N=6) | Escalation Cohort (MEDI4736 15 mg/kg Q3W) (N=7) | Exploration Durvalumab 20 mg/kg (Q4W) (N=21) | Expansion SCCHN Cohort (MEDI4736 10 mg/kg Q2W) (N=62) | Expansion Non-SCCHN HPV Positive Cohort (MEDI4736 10 mg/kg Q2W) (N=22) | Expansion NSCLC Cohort (MEDI4736 10 mg/kg Q2W) (N=304) | Expansion HCC Total Cohort (MEDI4736 10 mg/kg Q2W) (N=40) | Expansion ACM Cohort (MEDI4736 10 mg/kg Q2W) (N=21) | Expansion UM Cohort (MEDI4736 10 mg/kg Q2W) (N=24) | Expansion GEC Cohort (MEDI4736 10 mg/kg Q2W) (N=51) | Expansion TNBC Cohort (MEDI4736 10 mg/kg Q2W) (N=40) | Expansion PAC Cohort (MEDI4736 10 mg/kg Q2W) (N=31) | Expansion UC Cohort (MEDI4736 10 mg/kg Q2W) (N=201) | Expansion GBM Cohort (MEDI4736 10 mg/kg Q2W) (N=20) | Expansion OC Cohort (MEDI4736 10 mg/kg Q2W) (N=47) | Expansion STS Cohort (MEDI4736 10 mg/kg Q2W) (N=20) | Expansion SCLC Cohort (MEDI4736 10 mg/kg Q2W) (N=21) | Expansion MSI-high Cancer Cohort (MEDI4736 10 mg/kg Q2W) (N=62) | Expansion NPC Cohort (MEDI4736 10 mg/kg Q2W) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (11) | 5 (7) | 47 (74) | 5 (6) | 3 (12) | 1 (1) | 7 (20) | 2 (7) | 4 (7) | 43 (72) | 2 (2) | 10 (12) | 8 (14) | 5 (5) | 11 (22) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 1 (1) | 3 (4) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 12 (19) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 3 (3) | 29 (34) | 4 (4) | 3 (4) | 1 (1) | 2 (2) | 4 (5) | 5 (6) | 17 (21) | 2 (2) | 4 (4) | 2 (3) | 0 (0) | 6 (6) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 9 (10) | 5 (5) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 5 (6) | 4 (5) | 23 (28) | 11 (12) | 1 (2) | 4 (4) | 13 (27) | 2 (4) | 9 (12) | 20 (25) | 1 (1) | 15 (23) | 3 (5) | 3 (3) | 12 (24) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 7 (7) | 8 (11) | 0 (0) | 4 (4) | 4 (4) | 4 (5) | 1 (1) | 5 (5) | 3 (3) | 1 (5) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 10 (11) | 6 (7) | 48 (55) | 11 (12) | 4 (4) | 4 (4) | 16 (20) | 5 (5) | 9 (10) | 55 (63) | 2 (2) | 14 (16) | 3 (3) | 4 (4) | 13 (18) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 11 (18) | 6 (9) | 53 (96) | 10 (12) | 5 (8) | 5 (10) | 17 (19) | 5 (6) | 4 (5) | 36 (52) | 1 (2) | 11 (17) | 1 (1) | 0 (0) | 18 (37) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 17 (19) | 4 (4) | 1 (2) | 1 (1) | 5 (7) | 2 (2) | 4 (4) | 11 (14) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 10 (11) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 12 (12) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 15 (18) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 2 (6) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 3 (9) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 11 (13) | 2 (2) | 1 (1) | 1 (1) | 7 (18) | 2 (2) | 5 (5) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (6) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 12 (15) | 7 (8) | 67 (82) | 14 (16) | 5 (8) | 10 (14) | 13 (26) | 9 (9) | 10 (15) | 47 (70) | 5 (6) | 15 (25) | 2 (2) | 6 (6) | 18 (30) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 10 (13) | 6 (10) | 41 (53) | 10 (16) | 5 (5) | 4 (4) | 10 (35) | 7 (8) | 8 (16) | 27 (39) | 3 (4) | 10 (15) | 2 (3) | 4 (5) | 8 (15) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 2 (4) | 14 (16) | 6 (12) | 1 (1) | 5 (6) | 3 (3) | 5 (6) | 0 (0) | 26 (44) | 2 (2) | 4 (6) | 1 (1) | 1 (2) | 10 (12) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 13 (13) | 3 (3) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 6 (7) | 8 (10) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 3 (7) | 3 (5) | 8 (13) | 21 (29) | 11 (13) | 114 (165) | 20 (23) | 10 (10) | 9 (12) | 28 (73) | 7 (11) | 19 (24) | 73 (91) | 8 (8) | 19 (23) | 9 (11) | 6 (7) | 15 (19) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 17 (18) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (4) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 5 (6) | 1 (4) | 31 (42) | 11 (17) | 3 (3) | 2 (3) | 5 (5) | 6 (8) | 3 (3) | 28 (33) | 1 (1) | 9 (12) | 3 (3) | 2 (2) | 7 (11) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (11) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 9 (17) | 4 (6) | 33 (45) | 6 (18) | 4 (5) | 2 (3) | 7 (14) | 6 (6) | 4 (4) | 28 (34) | 3 (3) | 8 (8) | 5 (8) | 0 (0) | 11 (22) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (5) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 11 (12) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 8 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 9 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 25 (34) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (14) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 23 (29) | 1 (1) | 2 (2) | 4 (4) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 8 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (8) | 15 (17) | 4 (6) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 35 (55) | 0 (0) | 8 (8) | 4 (7) | 1 (2) | 10 (14) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (3) | 19 (25) | 9 (20) | 1 (2) | 1 (1) | 1 (1) | 4 (4) | 6 (14) | 17 (21) | 1 (1) | 7 (8) | 1 (2) | 0 (0) | 5 (9) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 20 (26) | 20 (30) | 2 (3) | 2 (2) | 3 (5) | 7 (12) | 5 (13) | 17 (21) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 5 (11) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 16 (21) | 9 (14) | 0 (0) | 4 (4) | 3 (3) | 4 (4) | 5 (12) | 11 (12) | 0 (0) | 4 (6) | 3 (4) | 0 (0) | 4 (8) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 8 (12) | 6 (8) | 1 (1) | 3 (6) | 1 (3) | 1 (3) | 2 (3) | 5 (8) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 12 (21) | 2 (2) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 21 (27) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Blood electrolytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (8) | 1 (1) | 12 (13) | 8 (10) | 0 (0) | 3 (5) | 3 (3) | 7 (11) | 7 (15) | 11 (14) | 0 (0) | 4 (7) | 2 (3) | 3 (3) | 4 (10) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 2 (3) | 24 (30) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 6 (8) | 16 (19) | 1 (1) | 9 (13) | 1 (3) | 2 (2) | 4 (7) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 9 (14) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 7 (9) | 7 (7) | 4 (7) | 80 (112) | 15 (17) | 6 (6) | 5 (5) | 22 (38) | 6 (6) | 11 (12) | 51 (60) | 4 (5) | 14 (17) | 2 (3) | 4 (4) | 10 (14) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (8) | 2 (2) | 18 (24) | 0 (0) | 4 (4) | 1 (1) | 8 (11) | 2 (2) | 5 (6) | 9 (12) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 4 (4) | 2 (3)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 16 (19) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (15) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (3) | 12 (15) | 4 (4) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 15 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 20 (22) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 22 (29) | 2 (4) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 11 (13) | 3 (3) | 4 (6) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 13 (17) | 3 (6) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 12 (15) | 0 (0) | 7 (8) | 0 (0) | 4 (5) | 4 (8) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 1 (1) | 31 (49) | 5 (8) | 0 (0) | 1 (3) | 5 (5) | 3 (5) | 3 (3) | 20 (25) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 4 (4) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (9) | 3 (3) | 44 (62) | 6 (6) | 9 (14) | 4 (5) | 1 (2) | 4 (5) | 3 (3) | 25 (40) | 1 (2) | 11 (15) | 5 (6) | 3 (3) | 9 (14) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 4 (4) | 49 (56) | 6 (6) | 3 (3) | 2 (5) | 13 (16) | 6 (6) | 8 (8) | 30 (44) | 2 (2) | 8 (8) | 4 (5) | 4 (4) | 14 (20) | 1 (2)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 10 (10) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 7 (10) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 8 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 25 (31) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 6 (9) | 1 (1) | 5 (8) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 1 (2) | 18 (23) | 6 (8) | 2 (2) | 2 (2) | 5 (33) | 2 (3) | 2 (2) | 16 (23) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 3 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 7 (8) | 1 (1) | 31 (41) | 3 (5) | 2 (2) | 5 (7) | 3 (3) | 4 (5) | 3 (4) | 14 (23) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 26 (32) | 3 (4) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 11 (15) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 0 (0) | 23 (24) | 6 (6) | 3 (4) | 2 (2) | 9 (22) | 4 (5) | 5 (5) | 11 (14) | 2 (3) | 5 (5) | 1 (1) | 3 (3) | 5 (9) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 8 (8) | 2 (3) | 33 (46) | 1 (1) | 2 (2) | 4 (5) | 5 (6) | 7 (8) | 7 (7) | 10 (15) | 9 (11) | 6 (7) | 2 (2) | 4 (4) | 9 (14) | 4 (5)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 2 (2) | 9 (10) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 6 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 16 (18) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 7 (7) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 8 (9) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 8 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 10 (10) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 24 (26) | 7 (7) | 1 (4) | 2 (6) | 13 (25) | 2 (2) | 1 (1) | 20 (22) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 7 (10) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (14) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (28) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (11) | 2 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (7) | 2 (2) | 9 (11) | 2 (2) | 77 (102) | 7 (8) | 4 (4) | 5 (6) | 12 (15) | 5 (5) | 8 (10) | 24 (27) | 2 (2) | 1 (2) | 2 (2) | 6 (7) | 10 (13) | 2 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 15 (21) | 5 (5) | 75 (100) | 8 (10) | 2 (2) | 6 (6) | 17 (22) | 10 (14) | 9 (10) | 27 (35) | 1 (1) | 9 (10) | 5 (5) | 3 (3) | 5 (5) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 8 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 24 (29) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (10) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 10 (13) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 4 (9) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 17 (20) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (2) | 14 (19) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 20 (23) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 10 (13) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 14 (15) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 7 (7) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 5 (15) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 2 (3) | 35 (49) | 16 (20) | 5 (7) | 4 (4) | 6 (8) | 5 (6) | 5 (8) | 15 (20) | 0 (0) | 7 (10) | 3 (3) | 0 (0) | 10 (12) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 2 (2) | 37 (54) | 5 (7) | 4 (7) | 7 (12) | 9 (13) | 1 (1) | 4 (6) | 23 (28) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 7 (13) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (13) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (16) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 7 (13) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT01693562/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT01693562/SAP_001.pdf